CLINICAL TRIAL: NCT04203602
Title: Assessment of Feasibility and Efficacy of Hospital Discharge Following Bariatric Surgery Using a Telepresence Robot: a Non-inferiority Randomized Controlled Trial
Brief Title: Hospital Discharge Following Bariatric Surgery by Telepresence Robot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Guilherme da Silva Mazzini, Principal Investigator, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25656919.4.0000.5327
Record Dates: First submitted 2019-12-13; First posted 2019-12-18 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Severe Obesity
Keywords: obesity; bariatric surgery
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Intervention Model Description: non-inferiority randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telepresence round (Experimental): Patients will be seen during ward rounds by the multidisciplinary team physically present, but with the surgeon remotely present via a telepresence robot.
  Interventions: Procedure: telepresence discharge
- conventional round (Active Comparator): Patients will be seen during ward rounds by the whole multidisciplinary team physically present, including the surgeon.
  Interventions: Other: Conventional discharge

INTERVENTIONS:
Procedure: telepresence discharge — Patients will be seen during ward rounds by the multidisciplinary team physically present, but with the surgeon remotely present via a telepresence robot.
  Arms: Telepresence round
Other: Conventional discharge — Patients will be seen during ward rounds by the whole multidisciplinary team physically present, including the surgeon.
  Arms: conventional round

SUMMARY:
This is a non-inferiority randomized controlled trial aimed to compare the effectiveness and feasibility of performing the ward round using a telepresence robot vs. a face-to-face ward round to discharge patients after bariatric surgery.

DETAILED DESCRIPTION:
This study is aimed to analyze the effectiveness and feasibility of performing the ward round using a telepresence robot (PadBot U, Inbot Technology Ltd, China), compared to the face-to-face ward round, for hospital discharge after bariatric surgery. Patients who underwent either laparoscopic Roux-en-Y gastric bypass or laparoscopic sleeve gastrectomy will be randomized to one of two groups: intervention group - who will be evaluated and discharged, on postoperative day (POD) 2, during ward rounds with the assistant team present, but the telepresent surgeon via robot; and control group - who will be evaluated and discharged, on POD 2, during ward rounds with the whole team physically present.

The study main hypothesis is that the ward rounds with the surgeon telepresent by a robot are not inferior to the face to face ward rounds, to evaluate and discharge patients after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients that underwent bariatric surgery (either laparoscopic Roux-en-Y gastric bypass or laparoscopic sleeve gastrectomy

Exclusion Criteria:

* complications during surgery; unable to sign informed consent; admitted to ICU; previous foregut surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-12-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Hospital discharges by robotic or face-to-face rounds | 2 days
  number of patients discharged on postoperative day 2 by robotic or face-to-face ward rounds

SECONDARY OUTCOMES:
contact with team | 2 weeks
  number of phone calls to the assistant team after discharge and before first visit at the clinic
complications, reoperations, readmissions | up to 30 days after surgery
  rates of early complications, reoperations, readmissions
Patients' and team's impressions | 2 days
  compare a validated questionnaire design to access patients' and team's impressions. There are 13 questions with answers valued from 1 to 5. The higher the score, the better the impression. The scores from the two groups are going to be compared in order to determine if patients' and team's impressions are similar with either robotic or face-to-face rounds.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme S Mazzini, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre; Cacio Wietzycoski, MD, Study Director — Hospital Unimed Vale do Caí
Locations (1):
- Unimed Vale do Caí, Montenegro, Rio Grande do Sul, Brazil